CLINICAL TRIAL: NCT00889265
Title: Prospective, Multi-Center Study of CopiOs® Pericardium Membrane With Puros® Cancellous Particulate Allograft for Localized Alveolar Ridge Augmentation
Brief Title: CopiOs® Pericardium Membrane for Localized Alveolar Ridge Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Collaborators: Zimmer Dental (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-801
Record Dates: First submitted 2009-04-26; First posted 2009-04-28 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Alveolar Ridge Defect
Keywords: Alveolar Bone Augmentation; Implant Surgery; Guided Bone Regeneration (GBR); Guided Tissue Regeneration (GTR); Bone Graft; Periodontal Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CopiOs Pericardium Membrane (Experimental): Subject's study site must exhibit a partially edentulous ridge of the maxilla or mandible with at least one tooth-span in length and less than 5.5mm in its smallest buccolingual dimension as measured by ridge-mapping calipers.
  Interventions: Device: CopiOs Pericardium Membrane

INTERVENTIONS:
Device: CopiOs Pericardium Membrane — CopiOs Pericardium, Puros Cancellous
  Other Names: Pericardium Membrane; Bovine Xenograft; Cancellous Particulate; Human Allograft

SUMMARY:
This is a prospective, multi-center study to evaluate the use of CopiOs Pericardium Membrane, a bovine xenograft, with use of Puros Cancellous Particulate Allograft, for the augmentation of localized alveolar ridge defects on either the maxilla or mandible.

DETAILED DESCRIPTION:
The study will evaluate the use of CopiOs Pericardium Membrane (CopiOs Pericardium), a bovine xenograft, with the use of Puros Cancellous Particulate Allograft (Puros Cancellous), a mineralized allograft, for the augmentation of localized alveolar ridge defects in edentulous sites. The purpose of the study will be to determine placement time, ease of use, stability, esthetics and to clinically evaluate the efficacy of the list products. A biopsy will be taken from a subset of the patient population, at one investigational site, to evaluate the grafted site's formation of new bone. The study hypothesis is that if CopiOs Pericardium and Puros Cancellous are used, the a single, localized alveolar ridge defect will clinically improve at an edentulous site.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of any ethnicity, between 18 and 99 years of age
* Health status of P1(ASA I) or P2 (ASA II), as classified by the American Academy of Anesthesiologists
* Able to communicate with the investigator and read, understand, and sign the informed consent form
* No evidence of active moderate or severe periodontitis
* Must be available for multiple follow-up visits for the duration of the study
* The study site must exhibit a partially edentulous ridge of the maxilla or mandible with at least one tooth-span in length and less than 5.5 mm in its smallest buccolingual dimension as measured by ridge-mapping calipers (#RIDGE-CALIPER, Salvin Dental Specialties, Inc., Charlotte, NC).

Exclusion Criteria:

* Inability or failure to maintain adequate oral hygiene
* Women who are bread-feeding, pregnant, or who intend to become pregnant during this study period. Women of childbearing potential should be practicing a medically accepted method of birth control
* Patients with unstable systemic diseases
* Patients with compromised immune system (e.g. uncontrolled diabetes, etc.) or unstable bleeding disorder
* Patients with active infectious diseases (e.g. hepatitis, tuberculosis, HEV, etc.)
* Patients with a mental disability that may hinder participation in the study (e.g. inability to follow through with oral hygiene instructions, postoperative instructions, follow-up commitments, etc.)
* Patients taking steroid medications or undergoing other immunosuppressive therapy
* Radiation, cancer therapy, and/or radiation specifically at the oral cavity within the last 6 months
* History of previous ridge augmentation at the site of interest
* Augmentation sites with localized pathology
* Patient who has participated in a clinical trial within 30 days of being enrolled in this study, is currently enrolled in another study, or plans to enroll in another study before the completion of of this study.
* Unresolved oral pathologies (e.g. periodontal disease, caries, etc.)
* Medications or conditions contraindicated for bone regeneration: methotrexate, corticosteroids, history of bisphosphonate use, cyclosporine-A, etc.
* Patients who have more than a minimal tobacco use (e.g. >10 cigarettes per day)
* Other conditions the investigator may feel would inhibit the patient from being a good candidate for this study or which are contraindicated in the Directions for Use.
* Note: Careful consideration should be given to alternative therapies prior to performing bone grafting in patients who have severe endocrine-induced bone diseases (e.g.hyperparathyroidism), or who are undergoing current therapy with drugs that intervene in calcium metabolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Mealy, Principal Investigator — University of Texas Health Sciences Center at San Antonio
Locations (4):
- United States (4):
  - University of Colorado Denver School of Dental Medicine, Aurora, Colorado
  - Indiana University, Indianapolis, Indiana
  - University of Texas Health Sciences Center at Houston, Houston, Texas
  - University of Texas Health Sciences Center at San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from June 2009 to February 2011. Subjects were recruited from patients attenting the PI's clinic and had one edentulous site which required lateral ridge augmentation prior to dental implant placement.
Pre-assignment Details: All enrolled participants took part in the study.
Groups:
- CopiOs Pericardium: Subject's study site must exhibit a partially edentulous ridge of the maxilla or mandible with at least one tooth-span in length and less than 5.5mm in its smallest buccolingual dimension as measured by ridge-mapping calipers.
  CopiOs Pericardium Membrane: CopiOs Pericardium Membrane (CopiOs Pericardium), a bovine xenograft 20mm x 30mm; Puros Cancellous Particulate Allograft (Puros Cancellous) 2 cubic centimeters (cc) of small particle (250-1000um).
Period: Overall Study
Arm/Group | CopiOs Pericardium
Started | 51 (Date Enrollment Started: 07/21/2009 Date Enrollment Completed: 02/15/2011 Total enrolled: 51)
Completed | 44
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 5
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | CopiOs Pericardium
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (15)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Change in Horizontal Ridge Widths From Baseline to 6 Months
Description: The primary outcome measure of the study was the average change in ridge width from baseline (pre operative/pre grafting) to 6 months post surgery. The ridge measurements were taken using ridge mapping calipers and recorded for each patient at baseline and 6 months. Baseline measurements were taken at the site of greatest ridge width deficiency as determined by the investigator and repeated at the same location for subsequent measurements. A radiographic template with a radiopaque foil was utilized to standardize clinical and radiographic measurements for each patient.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CopiOs Pericardium
Number analyzed (Participants) | 44
mm | 2.61 (1.8)

2. Secondary Outcome: Mean Wound Healing Index at 6 Months
Description: Score Description
  1. Uneventful wound healing with no gingival edema, erythema, suppuration, patient discomfort or flap dehiscence
  2. Uneventful wound healing with slight gingival edema, erythema, patient discomfort or flap dehiscence but no suppuration
  3. Poor wound healing with significant gingival edema, erythema, patient discomfort or flap dehiscence with suppuration
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CopiOs Pericardium
Number analyzed (Participants) | 42
units on a scale | 1.26 (0.44)

ADVERSE EVENTS:
Arm/Group | CopiOs Pericardium
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 14/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CopiOs Pericardium (N=51)
Graft not integrated, pain at surgical site (General disorders) | 5
Surgical Complications (Surgical and medical procedures) | 4
Infection at surgical site (Infections and infestations) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No